CLINICAL TRIAL: NCT02412137
Title: Effect of Compliance Counseling on Brace Success in Patients With Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Principal Investigator, Brandon Ramo, Principal Investigator, Texas Scottish Rite Hospital for Children
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112007-014
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counseled Patients (Experimental): The counseled cohort will have their brace wear compliance documented on the Brace Progress Report after the Orthotist downloads the time/temperature data onto a laptop from the sensor reader (A piece of computer hardware which the sensor clips into and is attached to the laptop via the USB port). The Orthotist will then reset the temperature logger discs and reinstall them into the padding in the inside front of the brace in order to monitor the next period of brace wear. This group will then be counseled for about 10 minutes or less regarding their brace-wear using the Brace Progress report as a checklist.
  Interventions: Other: Counseled cohort
- Non-counseled patients (Placebo Comparator): The non-counseled cohort will have their brace wear compliance documented on the Brace Progress Report after the Orthotist downloads the time/temperature data onto a laptop from the sensor reader (A piece of computer hardware which the sensor clips into and is attached to the laptop via the USB port). The Orthotist will then reset the temperature logger discs and reinstall them into the padding in the inside front of the brace in order to monitor the next period of brace wear. This group will not be counseled, and will only receive standard clinical care.
  Interventions: Other: Counseled cohort

INTERVENTIONS:
Other: Counseled cohort — This group will be counseled after brace temperature/date/time data is logged at each visit.

SUMMARY:
To measure the effectiveness of counseling on brace-wear compliance and curve progression in patients with adolescent idiopathic scoliosis. The investigators hypothesize that compliance is increased when it is measured and used to counsel patients, and therefore those patients will have less curve progression and fewer would need surgery.

A second purpose is to evaluate whether there is a correlation between BMI and brace effectiveness. Proposed theories for decreased effectiveness in patients with elevated BMI have included decreased compliance due to discomfort and decreased force exerted on the curve due to the larger habitus.

DETAILED DESCRIPTION:
The investigators plan to enroll 300 subjects prospectively with the hypothesis that some will be lost to followup, and would like a final number of at least 125 in each group. All patients who fit the inclusion criteria and consent to participate in the study will have two temperature monitors installed inside the padding in the front of their brace. The monitors will sample temperature every hour, with room temperature and body temperature representing periods of non-use and use respectively. Each temperature monitor is programmed to record temperature sequentially, so that a longer period of time can be monitored in case the patient's appointments get postponed beyond the time capacity of only one monitor. The monitors will be downloaded into a laptop computer by an orthotist in the scoliosis clinic each visit. A short questionnaire entitled the Brace Beliefs Questionnaire, consisting of 18 questions, will be administered to all patients at the time of brace prescription.

In approximately 50% of the patients, the information would be shared on each follow-up visit with the nurses, orthotist, and physician. Patients are not going to be randomized as communication in the clinic waiting room is common among braced patients. However, by having all patients treated by a specific physician included in either the counseling group, or if treated by a different physician in the standard care group, all patients in the waiting room at a given time would be enrolled in a single arm of the study. The patient and parent will then be given the visit's wear-time information and counseled regarding compliance using this information. A standardized progress report (Brace Progress Report) will be completed by the physician or orthotist.

In the other 50% of patients, only the person downloading the loggers would be aware of wear-time and that information would not be shared with the medical staff. Those patients will not receive detailed counseling regarding the actual hours of brace wear as documented by the temperature loggers, but instead will receive routine clinical care including a discussion about the importance of compliance. Radiographs routinely obtained in the clinic will be measured by the Principle Investigator. No extra radiographs will be obtained based on the participation in this study. The curve will be classified using the criteria of Lenke. Scoliosis will be measured by the Cobb angle technique and the Risser sign charted. Curve progression will be defined as progression of greater than or equal to six degrees. Patients with progression to greater than 45 degrees, who have surgery recommended, or who undergo spinal fusion surgery will be noted.

Enrollment and follow-up, gathering data, and analysis of that prospective data from 200 subjects is estimated to take approximately 5 years. We will not disclose to the subjects that information from the temperature monitors can be used to monitor compliance because such disclosure would change the purpose of the study.

With permission of the authors (Katz, et al, 2010) we will utilize de-identified BMI and brace compliance data from the 100 patients who completed their previous study. This data will be combined with the same information obtained from patient participation in this study since both studies essentially used the same method for measuring patient brace wear compliance. The increased numbers should lend stronger evidence to the findings. A target accrual number of 300 is expected (100 with de-identified retrospective data and 200 prospective study subjects).

SOURCES OF RESEARCH MATERIAL: Existing diagnostic data could come from the patients' medical records and radiographs, but temperature/date/time information downloaded from the loggers, data from the Brace Beliefs Questionnaire, and data recorded in the Brace Progress Report will be obtained specifically for research. Identifiable data obtained specifically for research purposes will be used to answer the study questions. Any data resulting from radiographic studies will be standard of care that is associated with the patient's clinical treatment, so no x-rays will be included for research purposes in this study.

The following information will be collected:

* Patient name/Identifier
* Age
* Gender
* Demographic information necessary to initiate contact with patient, including telephone numbers, address or language
* Date and results of physical exams from clinical records and radiographic studies
* Treatment history (surgical and non-surgical) and complications of treatment
* Temperature/date/time data downloaded from logger
* Data from short questionnaire (Brace Beliefs Questionnaire)
* Documentation of counseling session with patients who are in the counseling group using Brace Progress Report.
* Documentation of no counseling session in the "no counseling" group along with the amount of their brace wear compliance as recorded in the Brace Progress report.
* For the purpose of reporting any correlation between brace effectiveness and BMI, deidentified data from 100 patients previously enrolled in IRB#0598-2220 will be merged with the same data collected from physical exams and brace compliance data from this study.

RECRUITMENT OF SUBJECTS: Patients will be identified face-to-face as candidates for the study by the treating physician or orthotist at the scoliosis clinics at Texas Scottish Rite Hospital for Children as they present to clinic for diagnosis and treatment of their idiopathic scoliosis when the brace is initially prescribed. They will be invited, all study procedures will be explained to them, and they will be encouraged to have any questions answered. All patients will be informed that temperature loggers are going to be inserted in their orthoses, and that temperature information will be downloaded at each visit. Only the group that will receive counseling will be informed that the temperature information is a measure of brace compliance. The other group will not be informed that the temperature information indicates whether or not, and how often, the brace is worn. Informing them that the logger measures compliance would influence the outcome of the study, and therefore cannot be shared with the patients.

Study Procedures Screening Procedures Subjects will be identified and screened according to the inclusion/exclusion criteria as they present to clinic and are referred by their respective physicians to the Orthotics Department for bracing. This referral is standard clinical procedure.

Study Intervention After the study subject accepts the invitation to participate in the study, they will be asked to sign the consent documents and given copies for their records. The Research Coordinator will record documentation of the recruitment process, invitation to participate in the study, and informed consent on an Invitation Checklist. Subjects are routinely assigned randomly into one of seven orthopaedic physician's clinics on their first visit. Which of the two study groups they belong to will be determined by which physician is seeing them. All physician staff Orthopedists at TSRH have agreed to participate in this study and are listed as sub-investigators.The Principle Investigator will draw physician names to determine which ones will be receiving information about bracewear compliance that is downloaded from the monitors and then provide counseling to their patients, and which physician staff will not be receiving information about bracewear compliance at the patient visits, and thus will not be providing additional counseling based on this information. (1.One group will be counseled after brace temperature/date/time data is logged at each visit. 2. The other group will receive routine clinical care including a discussion about the importance of compliance.)

Procedures and Evaluations All subjects will be fitted by the Orthotist with a customized scoliosis brace that includes the two temperature logger discs (about the size of a nickel coin) which are fitted into the felt lining of the inside front of the brace. The subject will be given their first set of instructions regarding wear and care of the brace (standard clinical procedure) along with the Brace Beliefs Questionnaire (which should take less than 10 minutes and is being done specifically for research purposes. If the patient expresses anxiety at answering questions, they will asked whether they want to continue). At every subsequent clinic follow-up visit (see Follow-up below for frequency and duration), the counseling group will have their brace wear compliance documented on the Brace Progress Report after the Orthotist downloads the time/temperature data onto a laptop from the sensor reader (A piece of computer hardware which the sensor clips into and is attached to the laptop via the USB port). The Orthotist will then reset the temperature logger discs and reinstall them into the padding in the inside front of the brace in order to monitor the next period of brace wear. Depending on which group the patient has been assigned to, they will either be counseled for about 10 minutes or less regarding their brace-wear using the Brace Progress report as a checklist, or receive standard clinical care. Ideally, counseling would be done by the treating physician (standard clinical care) using the Bracing Progress Report Form (done for research purposes only). Counseling may also be done by nurse coordinators involved in the patient's care (which is standard clinical care) utilizing the same Bracing Progress Report Form if the treating physician is not available to do it. Data from the Brace Beliefs Questionnaire will be used to discover the subject's initial attitude about wearing the brace. Brace wear compliance data received from counseled patients will be compared to the same data received from the patients who have received standard clinical care to see whether counseling makes a difference in their compliance and thus their clinical outcomes.

Follow-up Patients will be followed for the duration of their bracing, which typically lasts approximately one to four years, and depends on the rate of their growth and curve progression. Data will be collected each time they present to clinic for follow-up, on average two to three times per year. Each patient will be followed until skeletally mature, two years following brace discontinuation, or until spinal fusion surgery is performed. Final outcomes (whether or not they progress to surgery) will be included in the data collected for this study.)

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of all races and ethnic backgrounds between the ages of 10 and 16, who have been or who are being treated for idiopathic scoliosis with a Boston brace at Texas Scottish Rite Hospital for Children. These patients will not have worn braces before and have scoliosis curves measuring from 25-45 degrees and are Risser 0, 1, or 2. Female patients will be premenarchal or <1 year post menarchal.

Exclusion Criteria:

* Patients with juvenile scoliosis (age less than 10 years), patients with non-idiopathic scoliosis, patients with curves measuring <25 degrees or >45 degrees at the time of brace prescription, patients previously treated with spinal surgery or orthoses, girls who are greater than one year postmenarchal, and patients who are Risser 3, 4, or 5.

Furthermore, if during the course of treatment a diagnosis of non-idiopathic scoliosis, i.e. if a spinal cord abnormality such as a syrinx, becomes apparent, the previously enrolled patient will be excluded from the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 245 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Karol, MD, Principal Investigator — Texas Scottish Rite Hospital for Children; Brandon Ramo, MD, Principal Investigator — Texas Scottish Rite Hospital for Children

REFERENCES:
- [Derived] Alvarez I, Poppino K, Karol L, McIntosh AL. Lack of in-brace x-rays in compliant AIS patients wearing full-time TLSO braces associates with failure. J Orthop Surg Res. 2021 Aug 31;16(1):540. doi: 10.1186/s13018-021-02650-9. PMID 34465348

RESULTS

PARTICIPANT FLOW:
Groups:
- Counseled Patients: The counseled cohort will have their brace wear compliance documented on the Brace Progress Report after the Orthotist downloads the time/temperature data onto a laptop from the sensor reader (A piece of computer hardware which the sensor clips into and is attached to the laptop via the USB port). The Orthotist will then reset the temperature logger discs and reinstall them into the padding in the inside front of the brace in order to monitor the next period of brace wear. This group will then be counseled for about 10 minutes or less regarding their brace-wear using the Brace Progress report as a checklist.
  Counseled cohort: This group will be counseled after brace temperature/date/time data is logged at each visit.
  144 patients were enrolled into this arm, 2 dropped out, 21 were lost to follow-up, 28 were excluded.
- Non-counseled Patients: The non-counseled cohort will have their brace wear compliance documented on the Brace Progress Report after the Orthotist downloads the time/temperature data onto a laptop from the sensor reader (A piece of computer hardware which the sensor clips into and is attached to the laptop via the USB port). The Orthotist will then reset the temperature logger discs and reinstall them into the padding in the inside front of the brace in order to monitor the next period of brace wear. This group will not be counseled, and will only receive standard clinical care.
  Counseled cohort: This group will be counseled after brace temperature/date/time data is logged at each visit.
  101 were enrolled into this arm, 9 were excluded, 14 were lost to follow-up.
Period: Overall Study
Arm/Group | Counseled Patients | Non-counseled Patients
Started | 144 | 101
Completed | 93 | 78
Not Completed | 51 | 23
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 21 | 14
Not completed — Physician Decision | 28 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Counseled Patients | Non-counseled Patients | Total
Number analyzed (Participants) | 144 | 101 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.52) | 14.1 (1.82) | 14.1 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 93 | 221
  Male | 16 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 144 | 101 | 245

OUTCOME MEASURES:

1. Primary Outcome: Brace Progress Report (i.e. Informing the Patient How Often They Were Wearing the Brace Versus Not Informing the Patient)
Description: Final treatment outcome of bracing vs surgery (i.e. how many patients had surgery versus no surgery for their spinal deformity). For each patient this time frame varies, patient "A" may effectively wear a brace that controls their spinal deformity for 4 years and never need surgical intervention, patient "B" may effectively wear a brace for a year but has a spinal deformity that continues to get larger and need surgical intervention, and patient "C" may wear a brace less than prescribed (noncompliant) for 2 years and progress to surgery.
Time Frame: up to 4 years, depending on length of bracing
Population: 144 patients were enrolled into the counseled patients arm, 2 dropped out, 21 were lost to follow-up, 28 were excluded. 101 were enrolled into the non-counseled arm, 9 were excluded, 14 were lost to follow-up.
Measure: Number; unit: participants
Arm/Group | Counseled Patients | Non-counseled Patients
Number analyzed (Participants) | 144 | 101
participants
  Completion Participants | 93 | 78
  Surgery: number analyzed (Participants) | 93 | 78
  Surgery | 26 | 29
  No Surgery: number analyzed (Participants) | 93 | 78
  No Surgery | 67 | 49

ADVERSE EVENTS:
Time Frame: Each patient was followed up to 4 years from initiation of the brace and skeletal maturity reached, bracewear that did not prevent curve progression requiring surgical intervention, or withdrawal from the project by either a) patient request, b) lost to follow-up or c) investigator exclusion.
Description: There were no adverse events to report.
Arm/Group | Counseled Patients | Non-counseled Patients
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/101
Other Adverse Events (participants affected / at risk) | 0/144 | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes